CLINICAL TRIAL: NCT02914990
Title: A Phase 1 Study of BPI-15086 in Patients With Epidermal Growth Factor Receptor T790M Mutation-positive Non-Small Cell Lung Cancer Who Have Progressed on Previous EGFR Tyrosine Kinase Inhibitor Therapy
Brief Title: Safety, Tolerability and Pharmacokinetic Profile of BPI-15086 in EGFR T790M Mutation-positive NSCLC Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTP-26511
Record Dates: First submitted 2016-09-20; First posted 2016-09-26 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BPI-15086 (Experimental): BPI-15086, orally administered daily
  Interventions: Drug: BPI-15086

INTERVENTIONS:
Drug: BPI-15086 — BPI-15086 is administered once daily with a starting dose of 25 mg in a 21-day cycle. When tolerated, increasing doses of BPI-15086 will be tested in subsequent cohorts, until a maximum tolerated dose is determined.

SUMMARY:
The main objective of this study is to evaluate the safety and tolerability of BPI-15086.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the safety and tolerability of BPI-15086. In addition, the anti-cancer effect of BPI-15086 in EGFR T790M mutation-positive advanced NSCLC patients who have progressed on a previous EGFR tyrosine kinase inhibitor therapy will also be evaluated. Biomarkers related to the efficacy of BPI-15086 will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, locally advanced or metastatic NSCLC patients, who is not suitable for surgery or radiotherapy
* Radiological documentation of disease progression while on a previous continuous EGFR TKI (e.g. icotinib, gefitinib, afatinib, neratinib, dacomitnib, or erlotinib) treatment
* Patients must fulfil one of the following:

  * Confirmation that the tumour harbours EGFR sensitivity mutation (exon 19 deletion, L858R and L861R, G719X)
  * Must have experienced clinical benefit from EGFR TKIs, according to the Jackman criteria
* Confirmation of T790M mutation positive after disease progression on EGFR TKIs
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 and estimated life expectancy of at least 12 weeks
* Measurable lesion per Response Evaluation Criteria in Solid Tumors(RECIST1.1)
* Adequate bone marrow, hepatic, and renal function
* Women: For pre-menopausal women who have a childbearing potential, they must have a pregnancy test within 7 days before starting treatment. The serum or urine pregnancy test must be negative and must be non-lacking; all patients (whether male or female) should be Adequate barrier contraceptive measures during the entire treatment period and 3 months after the end of treatment
* Have signed Informed Consent Form

Exclusion Criteria:

* Any other malignancy within 5 years of the first dose of study treatment
* Radiotherapy for target lesion within 4 weeks of the first dose of study treatment.
* From the treatment of reversible EGFR TKI drugs (e.g. Ectinib, Gefitinib, Erlotinib) to the first use of drugs, the time did not exceed 8 days or 5 half-lives (take the long time)；Irreversible EGFR TKI drugs (e.g. Alfatinib, Neratinib, Dacomitinib) did not last more than 14 days or 5 half-lives (take the long term)
* Investigational agents or anticancer drugs (Including cytotoxic chemotherapy) from a previous treatment regimen or clinical study within 14 days of the first dose of study treatment
* Prior treatment with other third generation EGFR TKIs, including osimertinib, rociletinib, EGF816, olmutinib, ASP8273 and avitinib
* Brain/meninges metastases unless asymptomatic, stable and not requiring steroids for at least 4 weeks prior to start of study treatment
* History of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease, radiological documentation of idiopathic pulmonary fibrosis at baseline; uncontrolled pleural effusion/pericardial effusion
* Any evidence of severe or uncontrolled systemic diseases, including CTCAE 2 or higher active infection, uncontrolled hypertension, unstable angina pectoris, congestive cardiac failure and severe liver/renal or metabolic disease
* Active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV)
* History of organ transplant; had surgery or severe injury within 4 weeks
* Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG eg, complete left bundle branch block, third degree heart block, second degree heart block, PR interval >240msec, or QRS> 110 msec
* Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval
* Poorly controlled hyperglycemia(fasting blood glucose level ≥7.0 mmol/L).
* Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment with the exception of alopecia
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of BPI-15086
* It is known that the study drug or any of its excipients (microcrystalline cellulose, lactose, crospovidone, hydroxypropyl cellulose, magnesium stearate) are severely allergic
* CYP3A4 strong inhibitors or inducers or Chinese herbal medicine for anti-tumor indications were used within 1 week before the first dose
* Abuse of drugs and medical, psychological or social conditions in patients may interfere with participating in the study or assessment of the results of the study
* Any condition that is unstable or may compromise patient safety and compliance with the study
* Researchers believe that patients who are not suitable for treatment with this regimen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Adverse events | 18 months
  Adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03

SECONDARY OUTCOMES:
Cmax | 4 weeks
Half life | 4 weeks
AUC | 4 weeks
Objective Response Rate | 12 weeks
Progression-Free Survival | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Department of Medical Oncology, Cancer Institute/Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No